CLINICAL TRIAL: NCT05893628
Title: Effect of Pectoralis Minor Length on Scapular Endurance and Core Endurance
Brief Title: Effect of Pectoralis Minor on Endurance
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assistant Prof., PhD, Selcuk University
Other Study IDs: 2023/05.25
Record Dates: First submitted 2023-05-25; First posted 2023-06-08 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pectoralis Minor Length
Keywords: pectoralis minor length; scapular muscle endurance; core muscle endurance; dominant arm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group
  Interventions: Other: muscle length and muscle endurance assessment

INTERVENTIONS:
Other: muscle length and muscle endurance assessment — Pectoralis Minor Length and muscle endurance evaluation

SUMMARY:
The aim of this study evaluate the effects of dominant and non-dominant pectoralis minor (PM) length on scapular and core muscle endurance in the absence of scapular dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* volunteered to participate in the study
* and did not have scapular dyskinesia according to the evaluations made

Exclusion Criteria:

* did not want to participate in the study
* and those with previous neurological or orthopedic upper extremity disorders,
* pain problems in any part of their body,
* previous abdominal surgery,
* and had communication problems

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adult women
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Pectoralis Minor Length and Index | 10 minutes
  PM length was measured with a caliper. The distance between the starting (origin) and ending (insertion) points of the PM muscle was measured, with the participant in supine position and the shoulder joint free.Pectoralis minor index (PMI) was obtained by dividing the PM length recorded in cm by the person's weight and multiplying the result by 100. PMI was determined by dividing the obtained value by weight
Scapular Dyskinesia | 15 minutes
  The lateral scapular slide test (LSST) was used to evaluate scapular dyskinesia. The distance between the inferior angle of the scapula and the closest vertebral spinous process in the standing upright position was bilaterally measured using a tape measure in three different positions
Scapular Muscle Endurance | 10 minutes
  Scapular muscle endurance was evaluated with the scapular isometric compression test. The participants were asked to stand upright with their arms on their sides and bring both shoulder blades closer together by maintaining this position as long as they could
Core Muscle Endurance | 15 minutes
  This evaluation was performed using McGill's torso muscular endurance test battery consisting of endurance tests in the trunk flexion, trunk extension (Sorensen), and right/left side bridge positions

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)